CLINICAL TRIAL: NCT05149352
Title: REStoring Mood After Early Life Trauma: the Effectiveness of Trauma-focused Therapy in Patients With Depression and Childhood Trauma
Brief Title: RESET-psychotherapy: the Effectiveness of Trauma-focused Therapy in Patients With Depression and Childhood Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting tot steun VCVGZ (Other); HSK Groep B.V. (Unknown); Altrecht (Other)
Responsible Party: Principal Investigator, Christiaan Vinkers, Prof. dr. mr. C.H. Vinkers, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL74405.029.20
Record Dates: First submitted 2021-11-02; First posted 2021-12-08 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder; Childhood Trauma
Keywords: Depression; Childhood trauma; Trauma-focused; Psychotherapy; Treatment; EMDR; Imagery rescripting
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment conditions. In one condition (control group) participants will receive a regular depression treatment that they would usually receive for their depression ('treatment as usual', TAU). In the other condition (intervention group) participants will receive trauma-focused therapy (TFT), additional and parallel to their depression treatment (TAU). In both treatment groups (TAU and TAU+TFT), treatment will be provided during a period of 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: As the interventions in these studies are psychotherapies, both participants and care providers cannot be masked from the treatment allocation. To ensure the objectivity of the research measures, the outcome assessors will be blinded to the allocated treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Active Comparator): Participants will receive an evidence-based psychotherapeutic intervention combined with/or pharmacotherapy (TAU)
  Interventions: Behavioral: Treatment as usual (TAU) for depression
- Treatment as usual (TAU) + Trauma-focused therapy (TFT) (Experimental): Participants will receive 6 to 10, 60-90 minute TFT sessions delivered over a period of 12 weeks, in addition to TAU.
  Interventions: Behavioral: Treatment as usual (TAU) for depression; Behavioral: Trauma-focused therapy (TFT)

INTERVENTIONS:
Behavioral: Treatment as usual (TAU) for depression — TAU for depression will be largely determined by the Dutch multidisciplinary practice guideline on depression (Spijker et al., 2013). This means that patients with CT-related depression will receive good clinical care, e.g. evidence-based psychotherapeutic interventions, such as cognitive behavioral therapy (CBT) or interpersonal therapy (IPT) combined with/or pharmacotherapy. Therapists who give TAU are not allowed to provide a trauma-focused intervention aimed at CT during the 12-week intervention period.
Behavioral: Trauma-focused therapy (TFT) — The content of TFT, delivered by another therapist than the therapist that will provide TAU, depends on the type of CT the patient reports. If the patient predominantly reports experiences of abuse, there are often clear memories of this abuse ('target images') present and Eye Movement Desensitization and Reprocessing (EMDR) is recommended as the treatment strategy. If the patient predominantly reports experiences of neglect, memories are often less identifiable, although these experiences can have a big impact on the development of maladaptive schemas. In this case, imagery rescripting (ImRs) is recommended as treatment strategy. If the patient reports both experiences of abuse and neglect, the therapist will discuss with the patient which type of CT has the greatest impact on the current depressive symptoms and starts with the indicated therapy. If indicated, the therapist can switch between EMDR and ImRs after a minimum of 4 sessions.
  Arms: Treatment as usual (TAU) + Trauma-focused therapy (TFT)

SUMMARY:
Depression is a debilitating psychiatric disorder with a recurrent and progressive course. Around 25% of depressive patients has experienced moderate to severe levels of childhood trauma (CT), resulting in earlier onset and more severe and recurrent depressions. There is currently no targeted treatment for CT-related depression. This is problematic as patients with CT-related depression respond poorly to standard depression treatments. The RESET-psychotherapy study proposes an innovative, targeted disease-modifying treatment strategy for CT-related depression. The main objective is to investigate the effectiveness of trauma-focused therapy (TFT), as an addition to regular depression treatment ('treatment as usual'; TAU), in reducing depression symptom severity in patients with CT-related depression. 158 adult patients will be randomized to receive a 12-week treatment with 1) TAU or 2) TFT in combination with TAU. The primary outcome measure is defined as depression symptom severity after 12 weeks treatment (post-treatment), measured with the Inventory of Depressive Symptomatology - Self Rated (IDS-SR).

DETAILED DESCRIPTION:
Depression is a debilitating psychiatric disorder with a recurrent and progressive course. Even though antidepressants and psychotherapy are often effective, a substantial proportion of patients does not respond to currently used evidence-based treatments. Around 25% of depressive patients has experienced moderate to severe levels of childhood trauma (CT), ranging from physical and emotional neglect to emotional, physical and sexual abuse. There is increasing evidence that depression related to childhood trauma (CT) is critically different from non-CT related depression: it emerges earlier in life with more severe and recurrent symptoms and has worse treatment outcomes. Therefore, there is a large and unmet need for novel therapeutic strategies for CT-related depression. Currently, there is no targeted treatment available for CT-related depression. Given the major role of trauma in CT-related depression, it is plausible that trauma-focused psychotherapies may be effective in this depression subtype. The current study aims to investigate the effectiveness of trauma-focused therapy (TFT), as an addition to 'treatment as usual' (TAU), in reducing depression symptom severity in patients with CT-related depression. It is expected that trauma-focused therapy will be a safe and rational strategy to enhance resilience and improve depression outcomes for patients with CT-related depression. RESET-psychotherapy is a 12-week randomized controlled clinical trial (single-blind RCT), in which TFT in combination with TAU will be compared to TAU only at various specialized mental healthcare units of mental health care institutions. The study population will consist of 158 adult patients who have a diagnosis of moderate to severe depression (according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)) and moderate to severe childhood trauma (CT). The primary outcome measure is defined as depression symptom severity after 12 weeks treatment (post-treatment), measured with the Inventory of Depressive Symptomatology - Self Rated (IDS-SR). Data will be collected during multiple assessments: at baseline (T0), after 6 weeks (T1), after 12 weeks (T2; post-treatment), and after 6 months post-treatment (follow-up, T3). Information about depressive symptoms, childhood trauma and other health-related outcomes will be assessed using self-report questionnaires and semi-structured clinical interviews. In addition, to better understand how and for who TFT works, stress-related biomarkers (hair cortisol, inflammatory and epigenetic biomarkers in the blood) will be examined pre- and post-treatment. A sub-group of patients (N=60, 30 per intervention group) will be asked to undergo fMRI scans pre- and post-treatment to measure stress-related brain activity (fMRI sub-study, ±60 minutes per fMRI session).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe depression, defined by a score ≥ 26 on the Inventory of Depressive Symptomatology - Self Rated (IDS-SR)
* DSM-5 diagnosis of MDD confirmed with the Dutch translation of the MINI-S for DSM-5
* Moderate to severe childhood trauma (CT) before the age of 18, defined by a score above validated cut-off on one or more of the following domains of the 28-item Childhood Trauma Questionnaire Short Form (CTQ-SF):

  * physical neglect: score ≥ 10
  * emotional neglect: score ≥ 15
  * sexual abuse: score ≥ 8
  * physical abuse: score ≥10
  * emotional abuse: score ≥ 13
* Sufficient mastery of Dutch language

Exclusion Criteria:

* Previous TFT on CT
* Other lifetime severe psychiatric comorbidity (bipolar disorder, psychotic disorder)
* Current alcohol/drug dependence
* Primary diagnosis of post-traumatic stress disorder (PTSD) or Acute Stress Disorder (ASD)
* Lifetime diagnosis of borderline personality disorder (BPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptom severity at post-treatment | Up to 12 weeks (post-treatment)
  Depressive symptom severity in patients with CT-related depression, measured with the Inventory of Depressive Symptomatology - Self Report (IDS-SR, with a total score ranging from 0 to 84, where higher scores indicate higher severity of depressive symptoms)

SECONDARY OUTCOMES:
Depressive symptom severity during treatment and at 9 months follow-up | Up to 9 months (follow-up)
  Depressive symptom severity in patients with CT-related depression, measured with the Inventory of Depressive Symptomatology - Self Report (IDS-SR, with a total score ranging from 0 to 84, where higher scores indicate higher severity of depressive symptoms)
Remission in CT-related depression | Up to 9 monts (follow-up)
  The presence or absence of DSM-5 Major Depressive Disorder (MDD), identified using the Major Depressive Disorder (MDD) section of the Dutch translation of the Mini International Neuropsychiatric Interview-Simplified (MINI-S).

OTHER OUTCOMES:
Functional disability | Up to 9 months (follow-up)
  General functioning and disability in major life domains, measured with the 12-item WHO Disability Schedule (WHODAS; with a total score ranging from 12 to 60, where higher scores indicate more disability or loss of function).
Anxiety symptoms | Up to 9 months (follow-up)
  The presence and severity of anxiety symptoms, determined with the Beck Anxiety Inventory (BAI; with a total score ranging from 0 to 63, where higher scores indicate higher severity of anxiety symptoms)
Insomnia | Up to 9 months (follow-up)
  Insomnia severity, measured with with the Insomnia Severity Index (ISI; with a total score ranging from 0-28, where higher scores indicate higher insomnia severity).
Subjective stress | Up to 9 months (follow-up)
  Subjective stress, determined with the Perceived Stress Scale (PSS; with a total score ranging from 0-40, where higher scores reflect greater perceived stress)
Suicidality | Up to 9 months (follow-up; if participants report suicidal ideation when completing the IDS-SR or undergoing the M.I.N.I. interview)
  The presence of suicidal ideation or behavior, determined with a shortened version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The suicidal ideation scale ranges from 0-5, where a score of 4 reflects an active suicidal ideation with some intent to act, but without a specific plan and a score of 5 reflects an active suicidal ideation with a specific plan and intent.
Hair cortisol (stress-related biomarker) | Up to 12 weeks (post-treatment)
  Long-term cortisol levels, assessed by hair samples collected pre - and post-treatment
Inflammatory markers (stress-related biomarkers) | Up to 12 weeks (post-treatment)
  Levels of C-reactive protein (CRP), Tumor Necrosis Factor-alpha (TNF-α) and Interleukin-6 (IL-6), assessed by blood samples drawn pre - and post-treatment
Epigenetic markers (stress-related biomarkers) | Up to 12 weeks (post-treatment)
  The DNA, extracted from blood samples drawn pre - and post-treatment, will be used for future exploratory epigenetic research. Epigenetic changes will be analyzed genome-wide using microarrays.
Brain structure - T1 (fMRI sub-study, not yet started, anticipated start April 2022) | Up to 12 weeks (post-treatment)
  A T1-weighted structural image will be acquired in order to obtain a high-resolution anatomic image of the brain with contrast between grey matter, white matter and CSF (cerebral spinal fluid).
Brain structure - DTI (fMRI sub-study, not yet started, anticipated start April 2022) | Up to 12 weeks (post-treatment)
  White matter (WM) tract integrity will be investigated by acquiring diffusion tensor images.
Functional dynamics of spontaneous neural activity (fMRI sub-study, not yet started, anticipated start April 2022) | Up to 12 weeks (post-treatment)
  Resting state fMRI (T2*-weighted echo planar images (EPIs), sensitive to blood oxygenation level-dependent (BOLD) contrast, will be obtained, covering the entire brain under rest)
Working memory (fMRI sub-study, not yet started, anticipated start April 2022) | Up to 12 weeks (post-treatment)
  Task-based fMRI** (T2*-weighted echo planar images (EPIs), sensitive to blood oxygenation level-dependent (BOLD) contrast, will be obtained, covering the entire brain under rest)
  ** Precise task to be determined; probably the n-back task or the digit-span task.
Emotion regulation (fMRI sub-study, not yet started, anticipated start April 2022) | Up to 12 weeks (post-treatment)
  Task-based fMRI (situation-focused volitional reappraisal task; T2*-weighted echo planar images (EPIs), sensitive to blood oxygenation level-dependent (BOLD) contrast, will be obtained, covering the entire brain)
Reward Processing (fMRI sub-study, not yet started, anticipated start April 2022) | Up to 12 weeks (post-treatment)
  Task-based fMRI (social incentive delay task; T2*-weighted echo planar images (EPIs), sensitive to blood oxygenation level-dependent (BOLD) contrast, will be obtained, covering the entire brain)

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan H Vinkers, Prof. dr., Principal Investigator — Amsterdam UMC, location VUmc and GGZ inGeest
Locations (3):
- Netherlands (3):
  - GGZ inGeest, Amsterdam, North Holland
  - HSK Groep, Woerden, Utrecht
  - Altrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol
Time Frame: Immediately following publication, no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] McLaughlin KA, Green JG, Gruber MJ, Sampson NA, Zaslavsky AM, Kessler RC. Childhood adversities and adult psychiatric disorders in the national comorbidity survey replication II: associations with persistence of DSM-IV disorders. Arch Gen Psychiatry. 2010 Feb;67(2):124-32. doi: 10.1001/archgenpsychiatry.2009.187. PMID 20124112
- [Background] Teicher MH, Samson JA. Childhood maltreatment and psychopathology: A case for ecophenotypic variants as clinically and neurobiologically distinct subtypes. Am J Psychiatry. 2013 Oct;170(10):1114-33. doi: 10.1176/appi.ajp.2013.12070957. PMID 23982148
- [Background] Nanni V, Uher R, Danese A. Childhood maltreatment predicts unfavorable course of illness and treatment outcome in depression: a meta-analysis. Am J Psychiatry. 2012 Feb;169(2):141-51. doi: 10.1176/appi.ajp.2011.11020335. PMID 22420036
- [Background] Spijker J, Bockting C, Meeuwissen J, Van Vliet I, Emmelkamp P, Hermens M, et al. Multidisciplinaire richtlijn Depressie (Derde revisie): Richtlijn voor de diagnostiek, behandeling en begeleiding van volwassen patiënten met een depressieve stoornis. Trimbos Instituut: Utrecht. 2013
- [Background] Driessen A., ten Broeke E. Schematherapie en EMDR gecombineerd bij complexe traumagerelateerde problematiek. Tijdschrift voor Gedragstherapie; 2014.
- [Derived] Gathier AW, Verhoeven JE, van Oppen PC, Penninx BWJH, Merkx MJM, Dingemanse P, Stehouwer KMKS, van den Bulck CMM, Vinkers CH. Design and rationale of the REStoring mood after early life trauma with psychotherapy (RESET-psychotherapy) study: a multicenter randomized controlled trial on the efficacy of adjunctive trauma-focused therapy (TFT) versus treatment as usual (TAU) for adult patients with major depressive disorder (MDD) and childhood trauma. BMC Psychiatry. 2023 Jan 17;23(1):41. doi: 10.1186/s12888-023-04518-0. PMID 36650502